CLINICAL TRIAL: NCT01841580
Title: Long-term Observation of Tear Proteomic Profiles and Ocular Surface in Trabeculectomy Patients Before and After Surgery
Brief Title: Proteomic Profiles in Trabeculectomy Patients
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Other Study IDs: R980/89/2012; 2013/020/A (Other: Singhealth Centralised Institutional Review Board)
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Glaucoma
Keywords: Tear proteins profiles; Longitudinal; Ocular surface damage; Trabeculectomy
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Approximately 70 million people world-wide are affected with glaucoma, of whom 6.7 million have bilateral blindness.5 Elevated intro-ocular pressure is the major modifiable risk factor in glaucoma, and reducing intraocular pressure to a consistently low level can delay disease progression and therefore, blindness.6 Topical intraocular pressure -lowering medication remains the first-line treatment for glaucoma, with surgical intervention playing a secondary role in cases suboptimally controlled with medication alone.

In this study, we plan to assess the change in tear proteins in trabeculectomy patients before and after operations. It is hoped that this study could help us gain more understanding of the possible mechanism accounting for the development of dry eye disease in glaucoma patients, which could help us develop better screening modalities and therapeutic agents for glaucoma patients at risk to prevent the development of dry eye disease.

DETAILED DESCRIPTION:
Study Objectives and Purpose

There are two primary aims in this study:

1. To assess changes in the tear proteomic profiles in pre-trabeculectomy and post-trabeculectomy patients
2. To assess the changes in clinical signs of the eye and tear film as well as dry eye symptoms.

Study Material Human Tears will be collected from patients in SNEC clinic

Study Design:

120 patients will be recruited for this study (details as described below). Schirmers I test, Tear Osmolarity, Tear Break Up Time (TBUT), Anterior segment optical coherence tomography (ASOCT) and Impression cytology will be done during the study visits. Subjective symptom and severity of dry eye disease will be assessed through Visual Analog Scale (VAS).

No. of visits:

There will be 4 visits in this study. Visit 1: Pre-trabeculectomy operation Visit 2: 6 month after trabeculectomy surgery Visit 3: 1 year after trabeculectomy surgery Visit 4: 3 years after trabeculectomy surgery

Selection and Withdrawal of Subjects Recruitment Criteria

1. 120 patients will be recruited from glaucoma clinics in SNEC
2. Patients age ≥ 21 years old
3. Patients who require trabeculectomy operation

Treatment of subjects

Study Procedures:

1. Fluorescein staining will be used to visualize patient eyes.
2. Schirmer's test will be used to measure the amount of tear production

   1. A small strip of filter paper will be inserted inside the lower eyelid
   2. A topical aneasthetic is placed into the eye before the filter paper to prevent tearing due to the irritation from the paper
   3. The eyes are closed for 5 minutes.
   4. The paper is then removed and the amount of moisture is measured
3. Impression cytology will be performed to collect the superficial conjunctival cells for analysis

   1. While the eye is still anaesthetized from Schirmer's test, one end of a filter paper will be impressed upon the temporal conjunctiva whilst the other hand is grasped in place with a blunt smooth edged forceps.
   2. The filter paper is removed from the conjunctiva with a peeling motion after 2-3 seconds.
   3. The paper is placed into an eppendorf tube for future analysis.
4. Tear osmolarity, Tear Break Up Time (TBUT) will be measured in all patients

   a) Tear osmolarity will be measured using the osmolarity chip, 3 chips per eye
5. Anterior segment optical coherence tomography will be performed to assess the tear meniscus and image for any conjunctivochalasis

   a) The patient will be asked to look at a target in the instrument while blinking normally. The instrument will scan the lower eyelid margin for imaging of the tear meniscus and conjunctivochalasis
6. Symptoms and severity of dry eye disease will be assessed through the Visual Analog Scale (VAS) system

Assessment of efficacy Outcome Measures

1. Symptoms and severity of dry eye disease will be quantified based on the Visual Analog Scale (VAS)11
2. Amount of moisture of the filter paper will be measured in Schirmer's test
3. Clinical assessment of dry eye disease through Tear break up time (TBUT) and Tear Osmolarity measurements
4. Tear meniscus height and area in the images obtained with optical coherence tomography

Target sample size 120 subjects will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. 120 patients will be recruited from glaucoma clinics in SNEC
2. Patients age ≥ 21 years old
3. Patients who require trabeculectomy operation

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients will be recruited for this study
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the tear protein profiles in trabeculectomy patients at 3 years | Baseline and 3 years

SECONDARY OUTCOMES:
Symptoms and severity of dry eye disease | Baseline and 3 years
Amount of tears will be measured | Baseline and 3 years
Tear Osmolarity will be measured | Baseline and 3 years
Tear meniscus height will be measured | Baseline and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre/ Singapore Eye Research Institute, Singapore, Singapore